CLINICAL TRIAL: NCT00093275
Title: A Phase II, Double-Blind, Placebo-Controlled, Multicenter Study to Assess the Efficacy and Safety of HP184 Administered Orally Once Daily for Twenty-Four Weeks in Adult Subjects With Chronic Spinal Cord Injury (CSCI)
Brief Title: HP184 in Chronic Spinal Cord Injury Subjects
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: ICD Study Director, sanofi-aventis
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DRI6213; HP184B/2002
Record Dates: First submitted 2004-10-05; First posted 2004-10-07 (Estimated); Last update posted 2008-08-21 (Estimated); Status verified 2008-08

CONDITIONS: Spinal Cord Injury
MeSH Terms: conditions — Spinal Cord Injuries

INTERVENTIONS:
Drug: HP184

SUMMARY:
The purpose of this study is to determine whether HP184 is effective in the treatment of chronic spinal cord injury (CSCI).

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects with incomplete (traumatic), chronic (defined as 18 months or more post spinal cord injury) SCI aged 18 to 65 years
* CSCI must be categorized in classes C or D in the ASIA impairment scale. (C = Incomplete impairment with motor function preserved below the neurological level, and more than half of key muscles below the neurological level have a muscle grade less than 3. D = Incomplete impairment with motor function preserved below the neurological level, and at least half of key muscles below the neurological level have a muscle grade more than or equal to 3).
* The level of the SCI must be between C4 and T10 (neurological)
* Subject has a measurable range of motion at the hips, knees and ankles and possesses potential propulsive activity (i.e. no functional contractures)
* Female subjects of childbearing potential (those who are not surgically sterile or who are less than 2 years postmenopausal) must be using two forms of birth control, including a primary and a secondary form and have a negative pregnancy test immediately prior to treatment. Primary forms of contraception include: tubal ligation, partner's vasectomy, intrauterine devices, birth control pills, and topical/injectable/implantable/insertable hormonal birth control products. Secondary forms of contraception include diaphragms, latex condoms and cervical caps; each must be used with a spermicide.

Exclusion Criteria:

* Any clinical evidence of recent fracture(s) within the last six months prior to study start.
* Any history of Multiple Sclerosis or peripheral demyelinating disease or neuromuscular disorder.
* Heart rate of less than 38 or greater than 100
* Ashworth spasticity score of 0/4 or 4/4 at the hip or knee.
* Subject whose medical condition requires mechanical ventilation.
* Lower motor neuron injury, such as those with conus medullaris or cauda equina injuries.
* Subject with lower extremity amputation or proximal femorectomy.
* Subject with pressure ulcers stages 3 and 4.
* Subject medically or mentally unstable in judgment of Investigator.
* Subject on tricyclic antidepressants such as nortriptyline, amitriptyline and imipramine.
* Subject with ASIA motor score of greater than or equal to 92.
* Subject with ASIA sensory score of greater than or equal to 200.
* Subject with history of seizure within 2 years prior to study start.
* Subjects who have participated in a clinical trial involving investigational medication within 30 days prior to administration of HP184 or placebo.
* Female subjects with positive urine pregnancy test.
* Female subjects who are breast feeding.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 262 (Actual)
Dates: Start 2004-10; Primary Completion 2005-12 (Actual); Study Completion 2005-12 (Actual)

PRIMARY OUTCOMES:
Change from baseline in total motor score of American Spinal Injury Association (ASIA) manual motor test at Week 24.

SECONDARY OUTCOMES:
Safety evaluation.

CONTACTS AND LOCATIONS:
Overall Officials: ICD CSD, Study Director — Sanofi
Locations (5):
- Sanofi-Aventis Administrative Office, Bridgewater, New Jersey, United States
- sanofi-aventis administrative Australia & New-Zealand administrative office, Macquarie Park, New South Wales, Australia
- Sanofi-Aventis Administrative Office, Berlin, Germany
- Sanofi-Aventis Administrative Office, Mumbai, India
- Sanofi-Aventis Administrative Office, Guildford Surrey, United Kingdom